CLINICAL TRIAL: NCT03345654
Title: Characterizing Variability in Hearing Aid Outcomes Among Older Adults
Brief Title: Individually-guided Hearing Aid Fitting
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Northwestern University
Other Study IDs: 1R01DC012289-06 (NIH)
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- New Hearing Aid Users fit with standard-of-care: Adults (18+) with hearing loss and newly fit with hearing aids
  Interventions: Other: Hearing Aids

INTERVENTIONS:
Other: Hearing Aids — The signal processing of newly fit hearing aids will be evaluated for acceptability based on the toolset, which takes additional patient information beyond hearing threshold (like cognition) to determine the optimal hearing aid signal processing strategies.
  Other Names: Hearing Aid Fitting

SUMMARY:
This translational project aims to optimize the fitting of hearing aids by development and clinical validation of a toolset that guides signal processing choice based on the individual auditory and cognitive abilities of the patient.

DETAILED DESCRIPTION:
The clinical trial portion of the project will validate clinical use of the toolset by evaluating a population of patients fit using current standard of care. Patient characteristics, such as audiological profile and cognition, will be collected. Their hearing aid settings will then be evaluated to determine if they meet toolset guidelines for signal processing based on their patient characteristics (auditory and cognition). Data regarding subjective and objective hearing aid outcomes will also be collected. It is hypothesized that hearing aid fittings that meet the standards of the proposed clinical toolset will result in better patient outcomes (objective and subjective) and fewer post-fitting visits.

ELIGIBILITY:
Inclusion Criteria:

* sensorineural hearing loss with pure-tone thresholds 70 dB HL or better at octave frequencies between 250 and 4000 Hz, 4 (.5, 1, 2, 3 kHz)
* frequency pure-tone average (PTA) of ≥ 30 dB HL.
* Listeners will have symmetrical losses, defined here as a 4-frequency PTA difference between ears ≤ 20 dB HL.

Exclusion Criteria:

* recent (within last 12 months) hearing aid use
* conductive loss (air-bone gaps > 10 dB at any frequency and/or abnormal immittance) -
* scoring < 23 on the Montreal Cognitive Assessment
* Hearing loss exceeding the limits that can be successfully aided with hearing aids (i.e., profound hearing loss)
* Hearing loss remediated with a cochlear implant (cannot wear hearing aids)
* Significant history of otologic or neurologic disorders
* Non English speaking participants
* Any clinically significant unstable or progressive medical condition
* Any condition which, in the opinion of the investigator, places the participant at unacceptable risk if he or she were to participate in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be recruited from the Northwestern University Center for Audiology, Speech, Learning, and Language. They will be adults (18+) who are new hearing aid users with no recent prior hearing aid experience. Any patient at the clinic who purchases a new pair of hearing aids and meets the study criteria will be provided information about the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Speech intelligibility | Baseline at initial fit, then post-intervention at final hearing aid appointment, about 30 days later
  Repeat low-context sentences

SECONDARY OUTCOMES:
Post-fitting adjustment visits | First 30 days of fitting
  Number of times hearing aid adjustments are made post-fitting
Speech and Spatial qualities questionnaire (SSQ) | Baseline at initial fit, then post intervention at final hearing aid appointment, about 30 days later
  Questionnaire evaluating subjective perception of hearing ability in different environments

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No